CLINICAL TRIAL: NCT03018054
Title: A Phase 2, Double-Blind, Parallel-Group, Placebo-Controlled Study of E6007 in Japanese Patients With Moderate Active Ulcerative Colitis
Brief Title: Study of E6007 in Japanese Patients With Moderate Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E6007-J081-201
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2018-07

CONDITIONS: Moderate Active Ulcerative Colitis
Keywords: moderate active ulcerative colitis; Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- E6007 30 mg (Experimental): Participants will receive E6007 30 milligrams (mg) once daily after breakfast.
  Interventions: Drug: E6007
- E6007 60 mg (Experimental): Participants will receive E6007 60 mg once daily after breakfast.
  Interventions: Drug: E6007
- Placebo (Placebo Comparator): Participants will receive matching placebo once daily after breakfast.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E6007 — once daily administration
  Arms: E6007 30 mg; E6007 60 mg
Drug: Placebo — once daily administration
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center study to evaluate the efficacy and safety of E6007 once daily for 8 weeks in Japanese participants with moderate active ulcerative colitis. Participants will be stratified by prior therapeutic treatment and Mayo score at Baseline, and will be randomized 1:1:1 to receive E6007 30 milligrams (mg), E6007 60 mg or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants aged from 20 to 74 years at the time of informed consent
* Participants with a diagnosis based on the Revised Diagnostic Criteria for Ulcerative Colitis (UC) issued by the Research Group for Intractable Inflammatory Bowel Disease Designated as Specified Disease by the Ministry of Health, Labor and Welfare of Japan (2013) at least 4 weeks before the start of administration of study drug
* Active UC participants as determined by Baseline complete Mayo score of 6 to 10 points with an endoscopic subscore of ≥2 and a rectal bleeding subscore of ≥1
* Participants who are currently being treated with oral 5-ASA or immunomodulator or corticosteroid with inadequate response or intolerance, or are corticosteroid dependent
* Participants being seen on an outpatient basis
* Has voluntarily consented, in writing, to participate in this study and is able and willing to comply with the requirements of this study protocol

Exclusion Criteria:

* Reduction in partial Mayo score of ≥3 points at Baseline from Screening
* Diagnosed with right-sided or segmental colitis, and proctitis from a Baseline endoscopy
* Received any anti-tumor necrosis factor (TNF) agent for over 2 years, or within 12 weeks prior to Baseline
* History of colectomy, or planning to have surgery for treatment of UC at Screening or Baseline
* White blood cell count below 3000/microliters (µL) at Screening
* History or suspected history of central nervous system disorder found at Screening or Baseline
* Current complication or suspected malignancy or toxic megacolon at Screening or Baseline
* Prior history or current complication of colonic dysplasia at Screening or Baseline
* History of any severe drug allergy at Screening or Baseline
* Received a live vaccine within 4 weeks prior to Baseline
* QTc repeatedly above 450 milliseconds (ms) on the electrocardiogram (ECG) test at Screening
* In the case of women: nursing mothers or pregnant women at Screening or Baseline
* Refusal to use medically suitable contraception (both the participant and the participant's partner) throughout the entire study period, if the participant is a man capable of reproduction or a woman of childbearing potential
* Female participants who want to become pregnant or male participants whose partners want to become pregnant throughout the entire study period
* Evidence of clinically significant disease that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments at Screening or Baseline
* History of any medical conditions or concomitant medical conditions that in the opinion of the investigator(s) would compromise the participant's ability to safely complete the study at Screening or Baseline
* A positive finding on the human immunodeficiency virus antigen and antibody test at Screening
* In tests conducted at Screening, a positive finding for any of the following: hepatitis B virus surface antigen, hepatitis B virus surface antibody, hepatitis B virus core antibody, or hepatitis C virus antibody
* Any result other than negative on the tuberculosis test at Screening
* Findings indicating a history of tuberculosis on chest X-ray during Screening
* History of drug or alcohol dependency or abuse within approximately the last 2 years prior to Screening or Baseline
* Use of illegal recreational drugs at Screening or Baseline
* Currently enrolled in another clinical trial or used any investigational drug or device within 16 weeks preceding informed consent

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Mayo score at 8 weeks | Baseline; 8 weeks

SECONDARY OUTCOMES:
Number of participants with abnormal, clinically significant laboratory values | up to 8 weeks
Change from Baseline in body temperature at 8 weeks | Baseline; 8 weeks
Change from Baseline in diastolic blood pressure and systolic blood pressure at 8 weeks | Baseline; 8 weeks
Change from Baseline in heart rate at 8 weeks | Baseline; 8 weeks
Change from Baseline in respiratory rate at 8 weeks | Baseline; 8 weeks
Change from Baseline in standard 12-lead electrocardiogram (ECG) values | Baseline; 8 weeks
Number of participants with abnormal, clinically significant chest X-ray findings | up to 8 weeks
Number of participants with any serious adverse event and number of participants with any non-serious adverse event | up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (64):
- Japan (64):
  - EA Pharma Trial Site #1, Nagakute, Aichi-ken
  - EA Pharma Trial Site #1, Nagoya, Aichi-ken
  - EA Pharma Trial Site #2, Nagoya, Aichi-ken
  - EA Pharma Trial Site #3, Nagoya, Aichi-ken
  - EA Pharma Trial Site #1, Toyoake, Aichi-ken
  - EA Pharma Trial Site #1, Toyota, Aichi-ken
  - EA Pharma Trial Site #1, Hirosaki, Aomori
  - EA Pharma Trial Site #2, Hirosaki, Aomori
  - EA Pharma Trial Site #1, Sakura, Chiba
  - EA Pharma Trial Site #1, Urayasu, Chiba
  - EA Pharma Trial Site #1, Matsuyama, Ehime
  - EA Pharma Trial Site #1, Ōgaki, Gifu
  - EA Pharma Trial Site #1, Takasaki, Gunma
  - EA Pharma Trial Site #1, Fukuyama, Hiroshima
  - EA Pharma Trial Site #1, Obihiro, Hokkaido
  - EA Pharma Trial Site #1, Sapporo, Hokkaido
  - EA Pharma Trial Site #2, Sapporo, Hokkaido
  - EA Pharma Trial Site #1, Nishinomiya, Hyōgo
  - EA Pharma Trial Site #1, Kanazawa, Ishikawa-ken
  - EA Pharma Trial Site #2, Kanazawa, Ishikawa-ken
  - EA Pharma Trial Site #1, Morioka, Iwate
  - EA Pharma Trial Site #1, Takamatsu, Kagawa-ken
  - EA Pharma Trial Site #2, Takamatsu, Kagawa-ken
  - EA Pharma Trial Site #1, Kamakura, Kanagawa
  - EA Pharma Trial Site #1, Kawasaki, Kanagawa
  - EA Pharma Trial Site #1, Sagamihara, Kanagawa
  - EA Pharma Trial Site #1, Yokohama, Kanagawa
  - EA Pharma Trial Site #1, Tsu, Mie-ken
  - EA Pharma Trial Site #1, Sendai, Miyagi
  - EA Pharma Trial Site #2, Sendai, Miyagi
  - EA Pharma Trial Site #1, Nagaoka, Niigata
  - EA Pharma Trial Site #1, Kurashiki, Okayama-ken
  - EA Pharma Trial Site #1, Sayama, Osaka
  - EA Pharma Trial Site #1, Suita, Osaka
  - EA Pharma Trial Site #1, Kawagoe, Saitama
  - EA Pharma Trial Site #1, Izumo, Shimane
  - EA Pharma Trial Site #1, Shimotsuga, Tochigi
  - EA Pharma Trial Site #1, Bunkyo, Tokyo
  - EA Pharma Trial Site #1, Chūō, Tokyo
  - EA Pharma Trial Site #1, Hachiōji, Tokyo
  - EA Pharma Trial Site #1, Minato, Tokyo
  - EA Pharma Trial Site #2, Minato, Tokyo
  - EA Pharma Trial Site #1, Mitaka, Tokyo
  - EA Pharma Trial Site #1, Shinagawa, Tokyo
  - EA Pharma Trial Site #1, Shinjuku, Tokyo
  - EA Pharma Trial Site #1, Ube, Yamaguchi
  - EA Pharma Trial Site #1, Kofu, Yamanashi
  - EA Pharma Trial Site #1, Chiba
  - EA Pharma Trial Site #1, Fukuoka
  - EA Pharma Trial Site #2, Fukuoka
  - EA Pharma Trial Site #1, Hiroshima
  - EA Pharma Trial Site #2, Hiroshima
  - EA Pharma Trial Site #1, Kagoshima
  - EA Pharma Trial Site #1, Kumamoto
  - EA Pharma Trial Site #1, Kyoto
  - EA Pharma Trial Site #2, Kyoto
  - EA Pharma Trial Site #1, Nagasaki
  - EA Pharma Trial Site #1, Niigata
  - EA Pharma Trial Site #1, Okayama
  - EA Pharma Trial Site #1, Osaka
  - EA Pharma Trial Site #2, Osaka
  - EA Pharma Trial Site #1, Saga
  - EA Pharma Trial Site #2, Saga
  - EA Pharma Trial Site #1, Toyama

IPD SHARING:
Plan to Share IPD: No